## **Participant Informed Consent Forms**

**Cultural Domain Analysis** 

CULTURAL DOMAIN ANALYSIS CONSENT FORM FOR PROJECT PARTICIPANTS Version 2 (10.06.2021)

Title of Project: Lamivudine (3TC) plus dolutegravir (DTG) dual therapy: a study on patients' experiences and perceptions

Name of Researcher and School: Giovanni Villa, Diego Garcia, and Caroline Ackley, BSMS

REC reference 21/NW/0070

| | | Please to Yes | ick box |
|---|---|---|---|
| | | Yes | No |
| • | I consent to being interviewed by the researcher | | |
| • | I agree to allowing the interview to be audio-recorded | | |
| • | I agree to allowing the digital notecards to be saved during the interview | | |
| • | I consent to the use of anonymised quotes in publications from the research | | |
| • | At this point in time I agree to be contacted again for a further interview or focus group discussion. If I change my mind, I will inform the researchers. | | |
| • | I understand that in exceptional circumstances e.g. where the health, welfare and safety of myself or others is compromised by information I might disclose, the researcher will be legally required to pass this information to your GP or the HIV clinical team. | | |
| • | I understand that any information I provide is confidential, and that no information that I disclose will lead to the identification of any individual in the reports on the project, either by the researcher or by any other party | | |
| • | I have read the information sheet, had the opportunity to ask questions and I understand the principles, procedures and possible risks involved. | | |

| data fo<br>such in | ent to the processing of my personal information and rethe purposes of this research study. I understand that formation will be treated as strictly confidential and d in accordance with the Data Protection Act 2018. |
|---|---|
| choose<br>can wit<br>penalis | stand that my participation is voluntary, that I can not to participate in part or all of the project, and that I hdraw at any stage of the project without being ed or disadvantaged in any way nor do I have to give s for this. |
| <ul> <li>I agree</li> </ul> | to take part in the above Brighton and Sussex Medical (BSMS) research project |
| Participant<br>Name:<br>Signature | |
| Date: | |
| Researcher<br>Name: | |
| Signature | |
| Date: | |